CLINICAL TRIAL: NCT02742116
Title: Evaluation of the Implementation of Expanded Carrier Screening Before Pregnancy in Hong Kong
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: The Family Planning Association of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: ECSFPA1.0
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Genetic Testing
Keywords: Expanded carrier screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva/swab shall be collected from patient/couple for Hereditary Disease DNA screening test by DrGene.
  Blood sample shall be taken by venipuncture of women for Fragile X carrier screening by Prenatal Diagnostic Laboratory, Tsan Yuk Hospital
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA screening before Pregnancy — Saliva/swab shall be collected from couple for Hereditary Disease DNA screening test. Blood sample shall be taken by venipuncture of women for Fragile X carrier screening A pre-test questionnaire will be conducted to assess subject's knowledge, views and preferences in receiving expanded carrier screening, choice of having concurrent or sequential screening, factors affecting their choices, anxiety level, and their willingness to pay for the test.
  A post-test self-administered questionnaire shall be filled in by the patient on receiving the test results.
  Couples who receive a screen positive result shall be subsequently referred to Queen Mary Hospital for joint counselling by clinical geneticist and gynaecologist. This consultation shall be audiotaped or videotaped.

SUMMARY:
The objectives are to:

1. Assess patient's views and preferences in receiving expanded carrier screening
2. Perform qualitative study on post testing counselling on screen positive individuals and at risk couples

DETAILED DESCRIPTION:
This study is to recruit 50 couples for Expanded carrier screening at Prepregnancy Checkup Clinic at the Family Planning Association.

Saliva swabs are collected from couples for Hereditary Disease DNA screening test by DrGene.

Blood samples are taken by venipuncture of women for Fragile X carrier screening by Prenatal Diagnostic Laboratory, Tsan Yuk Hospital.

A pre-test self-administered Questionnaire 1 will be administered to couples to assess their knowledge, views and preferences in receiving expanded carrier screening. This include collection of basic demographic information, answers to questions on basic principles of expanded carrier testing, reasons of having or declining the test, choice of having concurrent or sequential screening, factors affecting their choices, anxiety level of the patient is assessed by state-trait anxiety inventory. Their willingness to pay for the test is also assessed.

The test results will be available to couples in 6 week's time. A post-test self-administered questionnaire 2 will be administered to couples on receiving the test results at the clinic. These include assessment of anxiety level, any decision regret, outcome of test and resulting action.

The couples with a screen positive result will be referred to Queen Mary Hospital for a joint counselling by clinical geneticist and gynaecologist. This counselling/consultation shall be audiotaped or videotaped. The interviews will be transcribed verbatim. The data will be explored for themes and issues identified.

Statistics Questionnaire survey data shall be entered into SPSS. Descriptive statistics will be used to compare responses and choices of participants.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese couples who attend prepregnancy clinic
* Age 18 or above

Exclusion Criteria:

* Couples who cannot read or understand Chinese or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both female and male Chinese participants are being studied
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Patient acceptance and literacy of expanded carrier screening | 6 weeks
  Factors affecting the choice of expanded carrier screening in the prepregnancy and subfertility patients Identify counselling issues when expanded carrier screening is offered in the local setting

SECONDARY OUTCOMES:
Patient acceptance and literacy of expanded carrier screening | 6 months
  cost, false positives, workload generated from offering expanded carrier screening

CONTACTS AND LOCATIONS:
Overall Officials: Grace CY Wong, MD, Principal Investigator — The Family Planning Association of Hong Kong

IPD SHARING:
Plan to Share IPD: No